CLINICAL TRIAL: NCT05268497
Title: Assessment of Feasibility of Using Clinician-Directed Cognitive Behavior Therapy Supplemented by a Digital Application in Conjunction With Esketamine (SPRAVATO®) in Participants With Treatment-Resistant Depression
Brief Title: A Study to Assess Feasibility of Using Clinician-directed and Digital Application Supported Cognitive Behavior Therapy (CBT) in Conjunction With Esketamine in Participants With Treatment-resistant Depression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: due to budget decision and wanting to pursue other research priorities
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109113; NATRD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Esketamine; Cognitive Behavioral Therapy; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Esketamine (Experimental): Participants will receive esketamine nasal spray (Dose 1 or Dose 2) twice weekly for 4 weeks (Induction Phase), followed by once a week dose (Dose 1 or Dose 2) for 8 weeks (Maintenance Phase), in conjunction with an oral antidepressant. Clinician-directed cognitive behavioral therapy (CBT) supplemented with the Mindset app will be administered by a clinician following esketamine dosing once the participants is considered ready to engage in therapy, based on the clinician judgement of CBT readiness.
  Interventions: Drug: Esketamine; Behavioral: Cognitive Behavioral Therapy (CBT); Drug: Antidepressant

INTERVENTIONS:
Drug: Esketamine — Esketamine will be self-administered as nasal spray.
  Other Names: SPRAVATO; JNJ-54135419; Non-Investigational Medicinal Product/Auxiliary Medicinal Product (NIMP/AxMP)
Behavioral: Cognitive Behavioral Therapy (CBT) — Clinician-directed CBT supplemented by the Mindset app will be administered.
Drug: Antidepressant — Antidepressant will be administered orally.

SUMMARY:
The purpose of this study is to explore feasibility of combining clinician-directed cognitive behavioral therapy (CBT) supplemented with the Mindset app with esketamine therapy in participants with Treatment-resistant Depression.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. Any abnormalities must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must meet the Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) or recurrent MDD, without psychotic features, based upon clinical assessment confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Participant must have had nonresponse to greater than or equal to (>=) 2 different oral antidepressant treatments of adequate dose and duration in the current episode of depression
* Participant must be currently taking an oral antidepressant.
* Participant must be comfortable with self-administration of nasal spray medication and be able to follow the nasal spray administration instructions provided

Exclusion Criteria:

* Participant's depressive symptoms have previously demonstrated nonresponse to an adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar or related disorders (confirmed by the MINI), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before the start of the screening phase. A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary
* Participant has any anatomical or medical condition that, per the investigator's clinical judgment based on assessment, may impede delivery or absorption of nasal spray study drug
* Participant has known allergies, hypersensitivity, intolerance, or contraindications to esketamine/ketamine and/or its excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-07 (Estimated); Study Completion 2023-06-07 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) Scores (Participants) | Week 13
  The SUS provides a reliable tool for measuring the usability of a wide variety of products and services, including hardware, software, mobile devices, websites, and applications. It consists of a 10-item questionnaire with five response options for respondents; from strongly agree to strongly disagree.
Net Promoter Scale Scores (Participants) | Week 13
  Net promoter score is a market research measure that asks respondents to rate the likelihood that they would recommend a company, product, or a service to a friend or colleague. Responses are on a rating on a scale of 0 (not at all likely) to 10 (extremely likely).
Exit Survey | Week 13
  Exit survey is a survey including ratings regarding participant impression of features of the Mindset app.
Time Spent on Mindset App | From Week 2 up to Week 13
  Time spent on Mindset app will be reported for participants.
Number of Times Mindset App Used | From Week 2 up to Week 13
  Number of times the Mindset app is used will be reported.
Pattern of Mindset App Used | From Week 2 up to Week 13
  Pattern of Mindset app usage will be reported.
CBT Therapist Assessment of Completion of Action Plan | From Week 2 up to Week 13
  Assessment of completion of action plan will be done by CBT therapists through rating on a 5-point likert scale of the participant's progress.
Participant Interviews | Week 20
  Optional qualitative feedback from study participants (participant's interviews) on the usefulness of the Mindset in conjunction with esketamine will be reported.
SUS Scores (CBT Therapists) | Up to 14 months (at the end of study)
  The SUS provides a reliable tool for measuring the usability of a wide variety of products and services, including hardware, software, mobile devices, websites, and applications. It consists of a 10-item questionnaire with five response options for respondents; from strongly agree to strongly disagree.
Net Promoter Scale Scores (CBT Therapists) | Up to 14 months (at the end of study)
  Net promoter score is a market research measure that asks respondents to rate the likelihood that they would recommend a company, product, or a service to a friend or colleague. Responses are on a rating on a scale of 0 (not at all likely) to 10 (extremely likely).
Frequency of Use of Clinician Dashboard Used | From Week 2 up to Week 13
  Frequency of use of clinician dashboard will be reported.
Clinician Feedback | Up to 14 months
  Qualitative feedback on clinician dashboard and participant use of the mindset app in conjunction with esketamine (clinician feedback) will be reported.
Percentage of Participants Able to Engage in CBT | From Week 2 up to Week 13
  Percentage of participants able to engage in CBT on the day of dosing for each week of the study and overall will be reported.
Timing of CBT Readiness after Dosing | From Week 2 up to Week 13
  Timing of CBT readiness after dosing will be reported. Determination of readiness will be based on clinician judgement of CBT readiness to engage in CBT based on alertness and ability to concentrate after dosing.

SECONDARY OUTCOMES:
Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Scale Score | Pre-dose, 40 minutes and 90 minutes post-dose up to Week 4
  The MOAA/S will be used to measure treatment-emergent sedation with correlation to levels of sedation defined by the American Society of Anesthesiologists (ASA) continuum. The MOAA/S scores range from 0=no response to painful stimulus (corresponds to ASA continuum for general anesthesia) to 5=readily responds to name spoken in normal tone (awake; corresponds to ASA continuum for minimal sedation).
Clinician Administered Dissociative States Scale (CADSS) Score | Pre-dose, 40 minutes and 90 minutes post-dose up to Week 4
  The CADSS used to measure present-state dissociative symptoms, and to assess treatment-emergent dissociative symptoms. The CADSS consists of 23 subjective items, divided into 3 components: depersonalization (Items 3 to 7, 20, and 23), derealization (Items 1, 2, 8 to 13, 16 to 19, and 21) and amnesia (Items 14, 15, and 22). Participant's responses are coded on a 5-point scale (0=not at all through to 4=extremely). The total score is sum of the 23 items and range from 0 to 92, where 0 (best) and 92 (worst). A higher score indicates a more severe condition
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | From Week 2 up to Week 13
  Number of participants with TEAEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment
Number of Participants with Abnormalities in Vital Signs | From Week 2 up to Week 13
  Number of participants with abnormalities in vital signs (pulse/heart rate, blood pressure, and body temperature) will be reported.
Columbia Suicide Severity Rating (C-SSRS) Score | Up to Week 13
  C-SSRS is semi structured clinician-administered questionnaire designed to solicit the occurrence, severity, and frequency of suicide-related ideation and behaviors. The maximum score assigned for each participant will also be summarized into one of three categories: no suicidal ideation or behavior (0), suicidal ideation (1-5), suicidal behavior (6-10). Total score ranges from 1 to 10. Higher scores indicate greater severity.
Clinical Global Assessment of Discharge Readiness (CGADR) Score | From Week 2 up to Week 13
  The CGADR will be used to measure the participant's current clinical status and is the clinician's assessment of the readiness to be discharged from the study site. The clinician will answer "Yes" or "No" to the question "Is the participant considered ready to be discharged based on their overall clinical status (example, sedation, blood pressure, and other adverse events)?"

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Sheppard Pratt Health System, Baltimore, Maryland
  - University of Cincinnati, Dept of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency